CLINICAL TRIAL: NCT01474460
Title: Use of Phytonadione to Reduce INR Variability in Patients on Long-term Warfarin Therapy
Brief Title: Use of Phytonadione to Reduce International Normalized Ratio (INR) Variability in Patients on Long-term Warfarin Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James A. Haley Veterans Administration Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, To-Nga Huynh, PharmD., Anticoagulation Clinical Pharmacist, James A. Haley Veterans Administration Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000493
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Coagulation Delay
Keywords: warfarin; phytonadione; INR
MeSH Terms: interventions — Vitamin K 1; Vitamin K; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Placebo Comparator): The control group only receiving warfarin therapy (individualized therapy, hence no specific form, dosage, frequency and duration is applicable here - i.e. 5mg daily everyday for 6 months may be applicable to one patient but not all researched patients).
  Interventions: Dietary Supplement: phytonadione
- Phytonadione (Experimental): Patients receiving 200mcg of phytonadione.
  Interventions: Dietary Supplement: phytonadione

INTERVENTIONS:
Dietary Supplement: phytonadione — Phytonadione 200mcg PO daily for 6 months + normal dose of warfarin and standard of care treatment
  Other Names: Vitamin K; Coumadin

SUMMARY:
Background: Warfarin is used as an anti-coagulant in patients at risk of developing thrombosis. It has a narrow therapeutic index necessitating close monitoring of International Normalized Ratio (INR). According to a meta-analysis, patients were in therapeutic range only 63.6% of the time. This increases the risk of bleeding or thrombosis. Various retrospective and prospective studies have looked at supplementation with phytonadione in these patients to reduce the variability of INR showing an improvement in variability. Most of these studies have only been done in a small number of patients already on warfarin therapy. This study will focus on patients newly starting warfarin therapy.

Methods: This study is a prospective, randomized, controlled trial performed at James A. Haley Veterans' Hospital (JAHVA). Patients who meet criteria and sign informed consent will receive either phytonadione with warfarin or warfarin alone. Based on a power calculation for 80%, a total of 370 patients will be enrolled (185 participants in each arm). Participants will be randomized to either intervention or control. Intervention group participants will be prescribed their usual starting dose of warfarin along with 200 mcg phytonadione by mouth daily. Control group participants will be prescribed their usual starting dose of warfarin. Both groups will follow the usual standard of care. They will come in for a follow-up INR and warfarin dose titration at least once per week until therapeutic, and then as instructed up to every 6 weeks thereafter. Both groups will participate in anticoagulation clinic activities that constitute the current standard of care. Intervention will last for a total of 6 months for each participant once enrolled.

Hypothesis:Participants in the intervention group being supplemented with 200mcg of phytonadione will spend more total time with a therapeutic INR than participants in the control group.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* Be eighteen years of age and older
* Have a long-term indication for warfarin (will need to be on warfarin for 6 months or longer)
* Be a new patient on warfarin therapy, or a patient previously on warfarin therapy who has been taken off therapy for more than 2 weeks and needs to be titrated again
* Anticipate receiving medical care at the study site for the duration of the study
* Have transportation to and from the JAHVA
* Have read and signed the Informed Consent document after the study has been fully explained and has had all questions answered

Exclusion Criteria:

* Have liver or kidney failure
* Are on hemodialysis or peritoneal dialysis
* Are pregnant or planning to become pregnant
* Have Alzheimer's disease, cognitive impairment, or visual impairment
* Are not compliant with medications
* Are participating in another study
* Have scheduled surgery or are planning to undergo major surgery
* Cannot be reached by telephone
* Take over-the-counter vitamin K supplementation except multivitamins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2011-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study is to determine the length of time in therapeutic INR range for patients given phytonadione and warfarin compared to warfarin alone | 6 months

SECONDARY OUTCOMES:
Secondary outcomes include the number of adverse events in the form of bleeding or thrombosis for both groups. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: To-Nga Huynh, PharmD, Principal Investigator — James A. Haley VA Hospital
Locations (1):
- James A. Haley VA Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No